CLINICAL TRIAL: NCT05483374
Title: The Observational Clinical Registry of the European Reference Network on Rare Adult Solid Cancers: the Protocol for the Rare Head and Neck Cancers
Brief Title: The Head and Neck Registry of the European Reference Network on Rare Adult Solid Cancers
Acronym: EURACAN
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Associazione Italiana Oncologia Cervico Cefalica (Unknown); Ministry of Health, Italy (Other Government); European Union (Other); Alleanza Contro il Cancro (Other)
Responsible Party: Principal Investigator, Annalisa Trama, Head of the Epidemiology Valutative Unit, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: INT 43/21
Record Dates: First submitted 2022-07-11; First posted 2022-08-02 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer; Nasopharynx Cancer; Nasal Cavity and Paranasal Sinus Cancer; Salivary Gland Cancer; Middle Ear Carcinoma
Keywords: Rare cancers; head and neck cancers; registry; protocol
MeSH Terms: conditions — Head and Neck Neoplasms; Nasopharyngeal Neoplasms; Paranasal Sinus Neoplasms; Salivary Gland Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- epithelial tumours of nasal cavity and paranasal sinus: adult patients diagnosed with nasal cavity and paranasal sinus cancers (any stage of disease)
  Interventions: Other: observation
- epithelial tumours of nasopharynx: adult patients diagnosed with nasopharyngeal cancers (any stage of disease)
  Interventions: Other: observation
- minor and major salivary gland tumours: adult patients diagnosed with minor or major salivary gland cancers (any stage of disease)
  Interventions: Other: observation
- middel ear tumours: adult patients diagnosed with cancers of the middle ear (any stage of disease)
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — Not applicable, it is an observational registry

SUMMARY:
Cancer care for head and neck cancers is multidisciplinary and complex and knowledge on the rare ones is limited. There is a wide consensus that to support clinical research on rare cancers, clinical registries should be developed within networks specializing in rare cancers. Our hypothesis is that our head and neck cancer registry established in the framework of the European reference network on rare adults solid cancers will help to: describe the natural history of rare head and neck cancers; evaluate factors that influence prognosis; assess treatment effectiveness; measure indicators of quality of care.

The registry is a prospective observational real-world registry. It collects data from already available registries/database and/or directly from expert health care providers (HCP). Information are prospectively collected on patient characteristics; exposure, outcomes and potential confounders (https://euracan.eu/research/starter/rare-head-and-neck-cancer-registry/#codebook).

The registry if federated (i.e. data are stored by the data provider). Analyses will be performed using the federated learning approach which split computations into a local part and a central part. The data providers will share sub-computations only. Data quality checks are envisioned to assess whether data value are present, valid and believable. Validity and plausibility checks are embedded in the electronic case report form (CRF) in the form of alerts and errors during the data input. Additional checks are implemented in R and run using the federated learning to ensure a central data quality monitoring. The data analyses will include descriptive statistics showing frequency and patterns of patients' and cancers' variables; analytical analyses investigating the association of patients/disease and/or treatment characteristics and health outcomes.

Fondazione IRCCS Istituto Nazionale dei Tumori (INT) is the coordinator of the EURACAN registry as well as a data provider. At the INT, and at each HCP involved, responsible investigators ensure that the EURACAN registry will be implemented in compliance with the protocol, following the instructions and procedures described herein. Each HCP is a controller and will identify a data processor. The processing of patients' personal data taking part in the registry is compliant with local privacy legislation and the General Data Protection Regulation 2016/679 of the EU.

DETAILED DESCRIPTION:
Despite the rarity of each of the 198 identified rare cancers, collectively they represent 24% of all new cancer cases diagnosed in the EU28/yearly. Differences in survival for rare cancers exist across European countries suggesting the existence of inequalities in healthcare. Rare cancers in general get less scientific consideration and financial support than their more common counterparts. The generation of clinical evidence is more difficult due to the difficulties of conducting clinical trials for to the small number of patients and the paucity of accessible data, including data from cancer registries.

There is a wide consensus that to support clinical research on rare cancers, clinical registries should be developed within networks specializing in rare cancers. In the EU, a unique opportunity is provided by the European Reference Networks (ERNs). The ERNs are virtual networks of selected institutions targeting rare conditions. Three ERNs are dedicated to rare cancers: EuroBloodNet for rare haematological diseases, PaedCan for paediatric cancers and EURACAN for rare adult solid cancers ( https://euracan.eu/).

An EU-supported project Starting an Adult Rare Tumour Registry (STARTER) began on April 1st 2020 to develop the EURACAN registry. The registry initiated on the rare head and neck cancers including nasal cavity and paranasal sinuses (incidence rate 0.5/100,000), nasopharynx (incidence rate 0.5/100,000), salivary gland (incidence rate 1.5/100,000) and middle ear cancers (incidence rate 0.03/100,000), corresponding to 2,500, 2,500, about 8,000 and about 200 new cases/year in Europe, respectively (http://rarecarenet.istitutotumori.mi.it/analysis.php). Cancer care for head and neck cancers is complex in particular for the rare ones. Knowledge is limited, diseases are complex and often need multidisciplinary approach. Moreover, while most head and neck cancers are predominantly squamous cell carcinomas, salivary gland tumours include more than 20 distinct histological subtypes. Thus, heterogeneity add complexity to the rarity.

Against this background, the EURACAN registry on rare head and neck cancers was set up with the following objectives:

1. to help describe the natural history of rare head and neck cancers;
2. to evaluate factors that influence prognosis;
3. to assess treatment effectiveness;
4. to measure indicators of quality of care.

Furthermore, the registry aims to collect information, where available, on the storage of biological samples at the premises of the participating healthcare providers (HCPs). This will facilitate future studies on rare head and neck cancers biology.

The registry is designed to prospectively collect clinical data derived from diagnostic tests and treatments performed by the HCP as part of patient management. The data collected for the registry will not entail further examinations or admissions to the HCP and/or additional appointments to those normally provided. In other words, it will be an observational, real-world registry.

The registry will exploit data available from:

* national or regional registries/databases (DBs) dedicated to rare head and neck cancers (i.e. nasopharynx; nasal cavity and paranasal sinuses; salivary gland; and middle ear cancers)
* HCP registries/DBs;
* ad hoc data collection by HCPs.

The registry is federated thus, data are stored by the data provider. At the local level, data are pseudonymised.

The Personal Health Train (PHT) enables data from multiple organizations to be analysed without identifiable data leaving the organization. By keeping data at its source, no copies of datasets are generated and/or shared with third parties. Vantage6 is the open source implementation of the PHT (https://www.vantage6.ai). Vantage6 uses the mathematical principle of "federated learning" which is based on the mathematical principle of splitting computations into (a) parts at the station (local HCP or registry) and (b) a central part. The stations share sub-computations with the central server only. If federated learning does not work, the data, after quality validation, will be anonymised and sent to the coordination centre (i.e. National Cancer Institute of Milan [Fondazione IRCCS Istituto Nazionale dei Tumori, Milan-INT]).

Data analyses plan The data analyses will include descriptive statistics showing frequency and patterns of patients' and cancers' variables; analytical analyses investigating the association of patients/disease and/or treatment characteristics and health outcomes.

Descriptive statistics will be used to reconstruct the natural history of rare head and neck cancers (e.g. primary tumour growth rate and pattern, its metastatic dissemination, growth of metastases, association with other diseases etc.) and to report about quality of care.

Multivariable Cox's proportional hazards model and Hazard ratios (HR) for all-cause or cause specific mortality will be used to determine independent predictors of overall survival, recurrence and second primary cancer. Variables to include in the multivariable regression model will be selected based on the results of univariable analysis. The role of confounding of other covariates will be evaluated using stratified analysis or sensitivity analysis.

To assess treatment effectiveness, multivariable models, propensity score adjustment and progression-free survival will be performed.

High proportion of missing data threaten the validity of the inferences/prognostic models. Thus, a maximum of 10% of missing data will be allowed and missing data will be imputed using strategy such as unconditional/conditional mean or expectation maximum.

Sample size This is an observational clinical registry which implies a long-term data collection lasting until all the registry objectives are met. Being this registry an observational one, there won't be any tipe of sampling, therefore all the patients that meet the eligibility criteria will be selected. Only HCPs that treat at least 100 cases a year of all rare head and neck cancers are EURACAN member. As of April 2022, the registry is activating 10 HCPs and, with time, is envisioning to at least duplicate the number of data providers. Considering that we expected 6 centres in Italy, 2 centres in Germany, 1 centre in Czech Republic, 1 centre in Spain, 2 centres in France (400 cases per year)and the whole rare head and neck cases in The Netherlands (300 patients yearly, based on incidence estimations), we expect about 1700 patients with a rare head and neck cancer yearly.

Due to the observational nature of the registry, sample size justification is based on the precision of the estimates presented in terms of width of two-sided 95% Confidence Interval (CI) for a single proportion using the Simple Asymptotic method (in case of categorical variables) and in form of normal distribution for means (in case of continuous variables). Thus, for example, for a categorical endpoint (eg, proportion) a sample size of 80 patients (e.g. middle ear cases in 4 years) will achieve a maximum width of 95% CI on estimated proportions of 23.4% (i.e. estimated proportion +/- 11.7%). For continuous endpoints, a sample size of 80 patients will achieve a maximum width of 95% CI on estimated means of 0.46*SD (i.e. estimated mean +/- 0.23*SD, where SD=Standard Deviation).

For the analytical questions involving several different outputs and variables, it is not possible to define a summary of the sample size calculation. For this reason ad hoc analysis plans for each research question are envisioned.

Data quality checks Data quality checks aim to assess whether data value are present, valid and believable in terms of validity, plausibility and completeness. Validity and plausibility checks are embedded in the electronic case report form (CRF) in the form of alerts and errors during the data input. Additional checks are implemented in R. The R script, including the checks is downloaded locally from an online instruction repository. The R script extracts from the Research Electronic Data Capture (RedCap) (the IT solution used for the registry CRF) all the completed cases, stores a copy of the DB in the dedicated local server and runs the checks locally. The results of these checks are summarized in two reports: a summary and an individual report. Thanks to the Vantage6 software, the two reports (not the data) will reach the registry coordination team (INT) to be monitored and discussed with each data provider.

After the corrections made by the data providers, all checks will be re-run and quality reports reviewed by INT. Interaction with data providers will be reiterated until sufficient data quality is achieved. The DB with sufficient data quality will be saved and used for the federated learning analysis. These checks will be performed annually and will ensure high data quality within a federated DB.

Data to be collected Following the EURACAN registry objectives, data will be prospectively collected on patient characteristics, exposure and outcomes. Patient characteristics are descriptive patient data, such as patient demographics, including lifestyle, medical history, health status, etc. The registry will not collect genetic data. Exposure data focus on the disease, devices, procedures, treatments or services of interest. Outcome data describe patient outcomes (e.g. survival, progression, progression-free survival, death, etc.). In addition, data on potential confounders (e.g. comorbidity; functional status etc.) will be also collected (https://euracan.eu/research/starter/rare-head-and-neck-cancer-registry/#codebook).

Pitfalls There is a risk of limited representativeness due to the hospital-based nature of the registry and to the fact that hospital contributing to the registry are expert centres for these rare cancers. Representativeness of the registry will be tested comparing the registry data with population-based data in terms of relevant variables (eg. age, stage, prognosis). Adequate statistical (eg. marginal structural model) methods will be used if time-varying treatments/confounders and confounding by indication (selective prescribing) will be present, not to raise methodological problems.

Directed acyclic graphs can also be useful to identify the source of bias and will be utilized in the definitions of the path between covariates.

Clinical Follow-up could be an issue but active search of the life status of the patients will be guaranteed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epithelial tumours of nasopharynx; nasal cavity and paranasal sinuses; salivary gland cancer in large and small salivary glands; and middle ear (i.e. squamous carcinoma; adenocarcinoma; neuroendocrine; adenosquamous carcinoma, teratocarcinosarcoma, NUT carcinoma, odontogenic tumors) + neuroendocrine and adenocarcinoma in hypopharynx; oropharynx; larynx; oral cavity and lip + odontogenic carcinoma in oral cavity.
* Adult patients (aged ≥18 years).
* Diagnosis performed or verified by the expert centre entering the patient information in the registry.
* Patients entering the HCP at any clinical phase of the disease (diagnosis, treatment of primary cancer, treatment of recurrence, treatment of M+ etc.). The HCP can decide, based on its resources, the number of patients on whom it can collect data.
* New patients managed by the HCP from 2021 onwards plus patients managed by the HCP, who are actively followed up at the hospital, with year of diagnosis dating back to maximum 2018.

Exclusion Criteria:

• Patients (aged < 18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is an hospital based registry thus, hospitals experts in head and neck cancer.
  This registry won't select a sample of patients, but it will include every accordant patient present in each facility.
Sampling Method: Probability Sample
Enrollment: 13600 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive
Disease free survival | 1 year
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer.
The percentage of patients whose cancer shrinks or disappears after treatment. Treatment response expressed as a complete response; partial response; stable disease; progression based on clinical judgment on imaging. | 1 year
  A change related to treatment
Incidence of cancer treatment adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) | 1 year
  Any unexpected medical problem that happens during treatment with a drug or other therapy.
Percentage of patients with surgical complications as assessed by the Clavien-Dindo Classification | 1 year
  Any deviation from the ideal postoperative course that is not inherent in the procedure and does not comprise a failure to cure.
Percentage of patients treated according to clinical practice guidelines for head and neck cancer | 1 year
  Adherence to clinical practice guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Trama, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (12):
- Masaryk Memorial Cancer Institute, Brno, Brno, Czechia
- Assistance Publique-Hôpitaux de Paris - Hôpital Tenon, Paris, Paris, France
- University Hospital Essen, Essen, Hesse, Germany
- Italy (8):
  - IRCCS Ospedale Policlinico San Martino, Genova, Genova
  - IRCCS Ospedale San Raffaele, Milan, Milano
  - IRCCS Istituto Europeo di Oncologia, Milan, Milano
  - IRCCS Istituto Clinica Humanitas, Rozzano, Milano
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milan
  - Centro Nazionale di Adroterapia Oncologica, Pavia, Pavia
  - Nuovo Ospedale di Prato - S. Stefano, Prato, Prato
  - IRCCS Istituto Nazionale Tumori Regina Elena, Roma, Roma
- Fundacion Profesor Novoa Santos, A Coruña, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
The governance (link https://euracan.eu/registries/euracan-registry/registry-governance/)set the data access rules to the federated registry
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting in June 2022 and ending in January 2030
Access Criteria: 1. data remain the contributing HCPs or registries property and can't be moved
  2. each facility is free to access and use its own data for research
  3. each contributing facility can request access to the database adding a SC approved study protocol
  4. third parties proposing a research question should work with a EURACAN Principal Investigator (PI) and present a study protocol for SC review
  5. each EURACAN domain will define a domain registry working group to review the study protocols
  6. once approved, the scientific secretariat will ask the facility to confirm within 2 weeks if it wants to share its data. If it doesn't, it can opt out providing reason. If it doesn't answer, its data will not be used
  7. the scientific secretariat will inform the PI of the study about the SC decision
  8. the PI will arrange an ethical review that will be shared with the participating centers, which should respond within 60 days
  9. International collaboration of the EURACAN Registry is highly supported
URL: https://euracan.eu/registries/euracan-registry/head-and-neck-registry/

REFERENCES:
- [Background] Gatta G, Capocaccia R, Botta L, Mallone S, De Angelis R, Ardanaz E, Comber H, Dimitrova N, Leinonen MK, Siesling S, van der Zwan JM, Van Eycken L, Visser O, Zakelj MP, Anderson LA, Bella F, Kaire I, Otter R, Stiller CA, Trama A; RARECAREnet working group. Burden and centralised treatment in Europe of rare tumours: results of RARECAREnet-a population-based study. Lancet Oncol. 2017 Aug;18(8):1022-1039. doi: 10.1016/S1470-2045(17)30445-X. Epub 2017 Jul 4. PMID 28687376
- [Background] Gatta G, Trama A, Capocaccia R; RARECARENet Working Group. Epidemiology of rare cancers and inequalities in oncologic outcomes. Eur J Surg Oncol. 2019 Jan;45(1):3-11. doi: 10.1016/j.ejso.2017.08.018. Epub 2017 Sep 19. PMID 29032924
- [Background] Siesling S, Louwman WJ, Kwast A, van den Hurk C, O'Callaghan M, Rosso S, Zanetti R, Storm H, Comber H, Steliarova-Foucher E, Coebergh JW. Uses of cancer registries for public health and clinical research in Europe: Results of the European Network of Cancer Registries survey among 161 population-based cancer registries during 2010-2012. Eur J Cancer. 2015 Jun;51(9):1039-49. doi: 10.1016/j.ejca.2014.07.016. Epub 2014 Aug 15. PMID 25131265
- [Background] Trama A, Botta L, Foschi R, Visser O, Borras JM, Zagar T, Primic-Zakelj M, Bella F, Dimitrova N, Gatta G, Licitra L. Quality of Care Indicators for Head and Neck Cancers: The Experience of the European Project RARECAREnet. Front Oncol. 2019 Aug 28;9:837. doi: 10.3389/fonc.2019.00837. eCollection 2019. PMID 31555591
- [Background] Orlandi E, Alfieri S, Simon C, Trama A, Licitra L; RARECAREnet Working Group. Treatment challenges in and outside a network setting: Head and neck cancers. Eur J Surg Oncol. 2019 Jan;45(1):40-45. doi: 10.1016/j.ejso.2018.02.007. Epub 2018 Feb 14. PMID 29478741
- [Background] Gliklich RE, Dreyer NA, Leavy MB, editors. Registries for Evaluating Patient Outcomes: A User's Guide [Internet]. 3rd edition. Rockville (MD): Agency for Healthcare Research and Quality (US); 2014 Apr. Report No.: 13(14)-EHC111. Available from http://www.ncbi.nlm.nih.gov/books/NBK208616/ PMID 24945055
- [Derived] Trama A, Licitra L, Cavalieri S, Bonfarnuzzo S, Baili P, Ciarfella A, Parente P, Almadori G, Ansarin M, Bacigalupo A, Baumeister P, Baujat B, Bossi P, Cavalera E, Cercato MC, Dieleman F, Fakhry N, Ferraresi V, Gaino F, Galizia D, Halamkova J, Halme E, Hardillo J, Hofauer B, Kinloch E, Livi L, Locati LD, Mattheis S, Mercante G, Mirabile A, Molteni G, Orlandi E, Persio R, Sciallero S, Smeele L, Tagliabue M, Valentini V, Van Harpen C, Westphalen CB, Botta L. The observational clinical registry (cohort design) of the European Reference Network on Rare Adult Solid Cancers: The protocol for the rare head and neck cancers. PLoS One. 2023 Mar 16;18(3):e0283071. doi: 10.1371/journal.pone.0283071. eCollection 2023. PMID 36928072